CLINICAL TRIAL: NCT01777243
Title: A Single Dose First in Human Study of GSK2398852 Co-Administered With GSK2315698 in Patients With Systemic Amyloidosis
Brief Title: A Study to Evaluate the Safety of GSK2398852 When Co-administered With GSK2315698 in Patients With Systemic Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Imperial College London (Other); Heart Hospital (Unknown); Royal Free Hospital NHS Foundation Trust (Other); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115570
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Amyloidosis
Keywords: pharmacokinetic; systemic amyloidosis; safety; dose escalation; Carboxy Pyrrolidine Hexanoyl Pyrrolidine Carboxylate (CPHPC); biomarker; GSK2315698; GSK2398852; SAP; pharmacodynamic; co-administration; intravenous
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — miridesap

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A Arm (Experimental): Two subjects in Part A will receive starting dose level of GSK2398852 as 5 milligram (mg) [approximately equivalent to 0.1 mg/kilogram (kg)]. The next escalation dose levels in two subjects each are proposed as 1 mg/kg, 3 mg/kg, 10 mg/kg and 30 mg/kg. GSK2315698 will be administered at variable dosed until the concentration of the SAP mAb has fallen below 100 ng/mL.
  Interventions: Drug: GSK2398852; Drug: GSK2315698
- Part B Arm (Experimental): The precise selection of numbers of subjects and dose levels in Part B will be informed by the results from Part A.
  Interventions: Drug: GSK2398852; Drug: GSK2315698

INTERVENTIONS:
Drug: GSK2398852 — Unit dose strength: 100 mg/mL provided as 1 mL solution per vial. GSK2398852 dosage levels variable with the proposed starting dose level of GSK2398852 as 5 mg [approximately equivalent to 0.1 mg/ kg]. The next escalation dose levels are proposed as 1 mg/kg, 3 mg/kg, 10 mg/kg and 30 mg/kg.
Drug: GSK2315698 — Unit dose strength: 200 mg/mL stock to be diluted. GSK2315698 will be administered at variable dosed until the concentration of the serum amyloid P component monoclonal antibody (SAP mAb) has fallen below 100 ng/mL.

SUMMARY:
The study will be conducted in two parts. The first (Part A) will be an open label single dose escalation part beginning with the proposed starting dose level of GSK2398852 as 5 milligram (mg) [approximately equivalent to 0.1 mg/kilogram (kg)]. The next escalation dose levels are proposed as 1 mg/kg, 3 mg/kg, 10 mg/kg and 30 mg/kg. GSK2315698 will be administered at variable doses until the concentration of the serum amyloid P component monoclonal antibody (SAP mAb) has fallen below 100 nanogram/millilitre (ng/mL). Decisions about these next dose levels will be made following safety review of the prior subjects' data; dose levels may be changed (increased and lowered) and dose levels may be repeated depending on the observed safety such that Part A extension study may be performed. In addition, pharmacokinetics of GSK2315698 (SAP depleter) and GSK2398852 (anti-SAP mAb), and circulating SAP concentrations will be assessed. Dose escalation in Part A will continue to the highest well tolerated dose or the highest allowable dose. Subjects will be closely monitored and will undergo Equilibrium contrast Magnetic Resonance Imaging (EqMRI) including organ volume, Elastography and Liver Biopsy if required.

Part B will be a randomized partially blinded part with the principal objective of assessing the dose response of the GSK2398852 in more detail. Subjects will be assigned to one of approximately 5 dose groups from Part A. The precise selection of numbers of subjects and dose levels will be informed by the results from Part A.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been medically diagnosed with systemic amyloidosis and falls into one of the patient groups (small to moderate amyloid load involving the spleen for Part A; moderate to large amyloid load involving the spleen (to a moderate/large extent) for Part A (following agreement from external safety committee); moderate to large amyloid load involving the spleen and liver (spleen involved to a moderate/large extent) for Part A extension (if required); and moderate to large amyloid load involving the spleen (and liver in subset of subjects only) for Part B).
* Alanine aminotransferase (ALT) <3x upper limit of normal (ULN) and bilirubin <1.5x ULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* Subject is ambulant and capable of attending for the study visit schedule.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* A female subject is eligible to participate if she is of non-childbearing potential; or females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the approved contraception methods.
* Male subjects with female partners of child-bearing potential must agree to use one of the approved contraception methods.
* Smokers (<10 /day) are permitted but must be willing to abstain for the duration of residential study sessions

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* The subject has participated in a clinical trial and has received an investigational therapeutic product (unlicensed) within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). This timeframe will not apply to short term administration of GSK2315698 in study CPH114527.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* Estimated glomerular filtration rate (GFR)<30 milliliter (mL)/minute (min) [<60 mL/min for the first 4 subjects to be enrolled]
* Evidence of an active urinary sediment on microscopy as evidenced by the presence of red cell casts
* Decompensated cardiac failure or a recent history of syncope associated with cardiac disease.
* In a subject in whom there is a clinical suspicion of cardiac amyloid, an echocardiogram is consistent with significant cardiac amyloid, whether symptomatic or not.
* Clinically significant anaemia- hemoglobin (Hb) <9 gram (g)/deciliter (dL).
* Use of prohibited medications.
* Poor or unsuitable venous access.
* Subjects with a QT interval corrected using Fridericia's formulas (QTcF) of >480 ms or other electrocardiogram (ECG) abnormalities which, in the opinion of the investigator are clinically significant and may increase safety risk.
* Uncontrolled hypertension with systolic blood pressure (BP) >170 mmHg and /or diastolic >100 mmHg
* Presence of any co-morbid condition (e.g. severe or unstable coronary artery disease; moderate-severe chronic obstructive pulmonary disease) which in the opinion of the investigator would increase the potential risk to the subject.
* Subjects with active vasculitis
* Exclusions from Equilibrium contrast Magnetic Resonance Imaging (EqMRI) scanning [Contraindications to Magnetic Resonance Imaging (MRI) scanning including, but not limited to: Intracranial aneurism clips (except Sugita); History of intra-orbital metal fragments that have not been removed by an MD (as confirmed by orbital X-Ray); Pacemakers and non-MR compatible heart valves; Inner ear implants; History of claustrophobia; estimated GFR <30 mL/min (gadolinium exclusion)]
* Subjects with dementia or a diagnosis of cerebral amyloid angiopathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2015-12-22 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Safety of GSK2398852 as assessed by number of subjects with AEs in Part A and in Part B | Continuous throughout the study
  Adverse events (AEs) will be collected from the start of Study Treatment and until the follow-up contact.
Safety of GSK2398852 as assessed by clinical laboratory tests in Part A and in Part B | At scheduled intervals upto Day 42 in each Part.
  Safety data will include assessments of clinical laboratory tests (hematology, clinical chemistry and urinalysis).
Safety of GSK2398852 as assessed by vital signs measurements in Part A and in Part B | At scheduled intervals upto Day 42 in each Part.
  Safety data will include measurements of vital signs (semi supine systolic and diastolic blood pressure, pulse rate and temperature measured orally).
Safety of GSK2398852 as assessed by ECG readings in Part A and in Part B | At scheduled intervals upto Day 42 in each Part.
  Safety data will include single 12-lead electrocardiogram (ECG) readings obtained at each timepoint during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
PK profile of GSK2315698 and GSK2398852 in Part A and in Part B | In Part A and Part B on Day -2, Day 1 (pre-dose, 1 hour [hr], 2 hr, 3 hr, 4 hr, 8 hr, 12 hr), Day 2, Day 3, Day 4, Day 6, Day 14, Day 21, Day 42
  Pharmacokinetic (PK) profile GSK2315698 and GSK2398852 was performed to evaluate PK of single doses of GSK2398852 and GSK2315698 when co-administered.
Dose response of single doses of GSK2398852 when co-administered with GSK2315698 in Part B | Baseline, Day 6, Day 14 and Day 42 in Part B.
  The main measure of dose response will be determined by information from part A (and Part A extension if required). The options are: -Volume of distribution of gadolinium in the spleen as a measure of amyloid load (EqMRI); and -Liver histology examination for presence of giant cells, activation of macrophages, and amyloid clearance.

SECONDARY OUTCOMES:
SAP concentrations measurement | Baseline, Day -3, Day -2, Day -1, Day 42 in each Part.
  SAP concentrations before administration of GSK2398852 will be measured using Hycult ELISA assay; and SAP concentrations after administration of GSK2398852 will be measured by GSK assay in both Parts.
Measurement of anti-drug antibodies before and after treatment with GSK2398852 | Day 1 pre-dose, Day 21, Day 42 in each Part.
  Anti-drug antibodies before and after treatment with GSK2398852 will be measured to assess the immunogenicity of GSK2398852 when co-administered with GSK2315698.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Richards D, Millns H, Cookson L, Lukas MA. An observational, non-interventional study for the follow-up of patients with amyloidosis who received miridesap followed by dezamizumab in a phase 1 study. Orphanet J Rare Dis. 2022 Jul 9;17(1):259. doi: 10.1186/s13023-022-02405-7. PMID 35810311
- [Derived] Richards DB, Cookson LM, Barton SV, Liefaard L, Lane T, Hutt DF, Ritter JM, Fontana M, Moon JC, Gillmore JD, Wechalekar A, Hawkins PN, Pepys MB. Repeat doses of antibody to serum amyloid P component clear amyloid deposits in patients with systemic amyloidosis. Sci Transl Med. 2018 Jan 3;10(422):eaan3128. doi: 10.1126/scitranslmed.aan3128. PMID 29298867
- [Derived] Richards DB, Cookson LM, Berges AC, Barton SV, Lane T, Ritter JM, Fontana M, Moon JC, Pinzani M, Gillmore JD, Hawkins PN, Pepys MB. Therapeutic Clearance of Amyloid by Antibodies to Serum Amyloid P Component. N Engl J Med. 2015 Sep 17;373(12):1106-14. doi: 10.1056/NEJMoa1504942. Epub 2015 Jul 15. PMID 26176329
- See also: Results for study 115570 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115570?search=study&b'study_ids=115570'#rs